CLINICAL TRIAL: NCT03364465
Title: Effect of Lung Protective One-lung Ventilation With Fix and Variable Tidal Volume on Oxygenation and Outcome: Randomized, Controlled Trial
Brief Title: Lung Protective One-lung Ventilation With Fix and Variable Tidal Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Debrecen (Other)
Responsible Party: Principal Investigator, Tamas Vegh, MD, Head, Division of General, Vascular and Thoracic Anesthesia, University of Debrecen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DE RKEB/IKEB 4737-2017
Record Dates: First submitted 2017-11-22; First posted 2017-12-06 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Hypoxemia; Pulmonary Sepsis; ARDS, Human; Pneumonia
MeSH Terms: conditions — Hypoxia; Respiratory Distress Syndrome; Pneumonia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GruopFix (No Intervention): one-lung ventilation with constant tidal volume
- GroupVariable (Active Comparator): one-lung ventilation with variable tidal volume Intervention: change of ventilatory settings
  Interventions: Other: change of ventilatory settings

INTERVENTIONS:
Other: change of ventilatory settings — change of tidal volume during one-lung ventilation
  Arms: GroupVariable

SUMMARY:
During One-lung ventilation, the use of lower tidal volumes (VT) is helpful to avoid over-distension, provide sufficient oxygenation, but can result in increased atelectasis.

Nevertheless, it is not known if, during one-lung ventilation with constant low VT, moderate levels of PEEP combined with lung recruitment maneuvers are superior to variable low tidal volume for intraoperative oxygenation and protection against PPCs.

Aim of the study is to compare a strategy using constant tidal volume with recruitment maneuvers versus variable tidal volume with recruitment maneuvers during thoracic surgery in adults.

We hypothesize that in adult, non-obese patients undergoing thoracic surgery under standardized OLV with variable tidal volumes, modearte PEEP and recruitment maneuvers as compared to constant without recruitment maneuvers prevent PPCs.

Patients will be randomly assigned to one of two groups:

FIX TIDAL VOLUME GROUP (Groupfix): mechanical ventilation with constant (6 ml/kgIBW) tidal volume and PEEP of 5 cmH2O with recruitment maneuvers

VARIABLE TIDAL VOLUME GROUP (Groupvar): mechanical ventilation with variable (6 ml/kgIBW ± 33%) tidal volume with variable respiratory rate to maintain constant minute ventilation and PEEP of 5 cmH2O with recruitment maneuvers.

DETAILED DESCRIPTION:
Lung separation will be performed by DLT technique. Mechanical ventilation will be applied in volume-controlled mode. During two-lung ventilation, VT will be set at 8 mL/kg predicted body weight. During one-lung ventilation, in GroupFix VT will be decreased to 6 mL/kg PBW with 5 cmH2O PEEP.

In GroupVar VT will be 6 ml/kg predicted body weight ±33% with 5 cmH2O PEEP. Respiratory rate will be adjusted to maintain same minute ventilation as during two-lung ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for open thoracic or video-assisted thoracoscopic surgery under general anesthesia requiring OLV (no emergency surgery)
* BMI < 35 kg/m2
* Age ≥ 18 years
* Expected duration of surgery > 60 min
* Expected duration of anesthesia > 90 min

Exclusion Criteria:

* COPD GOLD 3+4, lung fibrosis, documented bullae, severe emphysema, pneumothorax
* uncontrolled asthma
* NYHA 3+4, CCS 3+4
* previous thoracic surgery
* ARDS (Berlin definition)
* documented pulmonary arterial hypertension > 40 mmHg syst
* documented or suspected neuromuscular disease (thymoma, myasthenia)
* planned mechanical ventilation after surgery
* bilateral procedures
* lung separation with other method than DLT (eg diff. airway, tracheostomy)
* surgery in prone position
* persistent hemodynamic instability, intractable shock
* intracranial injury or tumor
* enrollment in other interventional study or refusal of informed consent
* pregnancy (excluded by anamnesis and/or laboratory analysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
intraoperative oxygenation | 1 day
  PaO2 < 60 mmHg

SECONDARY OUTCOMES:
postoperative pulmonary complications | 90 days
  infiltrate on chest X-ray, fever, laboratory and physical signs of infection
postoperative extra-pulmonary complications | 90 days
  new atrial fibrillation
30-day survival/mortality | 30 days
  number of death within 30 days after surgery
90-day survival/mortality | 90 days
  number of death death within 90 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Debrecen, Department of Anesthesiology and Intensive Care, Debrecen, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Szamos K, Balla B, Paloczi B, Enyedi A, Sessler DI, Fulesdi B, Vegh T. One-lung ventilation with fixed and variable tidal volumes on oxygenation and pulmonary outcomes: A randomized trial. J Clin Anesth. 2024 Aug;95:111465. doi: 10.1016/j.jclinane.2024.111465. Epub 2024 Apr 6. PMID 38581926